CLINICAL TRIAL: NCT07094022
Title: A Randomized, Double-blind, Placebo-controlled, Single Center Study to Evaluate of the Improvement and Safety of Nutrilite Protein MetX Pro on Weight Management in Overweight Individuals With Dyslipidemia
Brief Title: Improvement and Safety of Nutrilite Protein MetX Pro on Weight Management in Overweight Individuals With Dyslipidemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amway (China) R&D Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 23-RD-08-AY-001
Record Dates: First submitted 2025-07-22; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Dyslipidemia; Obesity &Amp; Overweight
Keywords: High-protein Compound Beverages; Nutrilite Protein MetX pro
MeSH Terms: conditions — Dyslipidemias; Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrilite Protein MetX Pro (Active Comparator): Nutrilite protein MetX pro, 460g per pack. Ingredients: Mung bean protein, chickpea protein, isomaltulose, rice (glutinous rice) protein, green apple concentrated juice powder, inulin, xanthan gum, guar gum, silicon dioxide, food flavoring.
  Interventions: Dietary Supplement: Nutrilite Protein MetX Pro
- Placebo Product (Placebo Comparator): Placebo product , 460g per pack. Ingredient: Maltodextrin.
  Interventions: Dietary Supplement: Placebo Product

INTERVENTIONS:
Dietary Supplement: Nutrilite Protein MetX Pro — A total of 4 cans (460 g/can) of study products (Nutrilite Protein MetX Pro) are distributed to each participant. Participants need to take 16g each time, twice a day, for 4 weeks.
  Arms: Nutrilite Protein MetX Pro
Dietary Supplement: Placebo Product — A total of 4 cans (460 g/can) of placebo products are distributed to each participant. Participants need to take 16g each time, twice a day, for 4 weeks.
  Arms: Placebo Product

SUMMARY:
The goal of this randomized, double-blind, placebo-controlled, single center study is to evaluate the impact of Nutrilite Protein MetX Pro (the study product, a high-protein compound beverages supplemented with multiple plant proteins and apple extracts) on lipid profiles in the blood test in overweight individuals with dyslipidemia. The main question it aims to answer is:

- Does the intake of the study product improve the blood lipid profiles (TC,TG, LDL-C ) in terms of of overweight individuals with dyslipidemia?

Researchers will compare the product group to a placebo group to see whether the blood lipid profile is significantly better improved for participants in the product group.

Participants will:

* take randomly assigned products 16g/each time, twice a day for 4 weeks
* make four times site visits, once a week. Blood samples are collected for each visit, and Feces are collected for the first and last site visit.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years old
* Overweight or obese participants, 40 with a BMI of 24-28 kg/m², and 40 participants with a BMI greater than 28. The percentage of male participants is ≥40%. And the lipid profile with the following characteristics:
* TC (Total Cholesterol): 5.18-6.21 mmol/L;
* TG(Triglyceride): 1.70-2.25 mmol/L;
* LDL-C(Low-Density Lipoprotein Cholesterol): ≥ 3.4 mmol/L;
* Agree to sign the informed consent form.

Exclusion Criteria:

* Pregnant or lactating women, those with allergic constitutions, or those allergic to this test sample.
* Patients with severe diseases of the heart, liver, kidneys and hematopoietic system, as well as those with mental illness.
* Those who have taken lipid-lowering drugs or the like in the past two weeks, which has affected their judgment of the results.
* Patients with hyperlipidemia.
* The researcher determined that the participant was not suitable for this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2025-03-16 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
Lipid profile index-TC | baseline day 0, day 28
  TC (Total Cholesterol) concentration level in the blood sample test: normal range 3-5.2 mmol/L; higher than 5.2 mmol/L is abnormal.
Lipid profile index-TG | baseline day 0, day 28
  TG (Triglyceride) concentration level in the blood sample test : normal range 0~1.7 mmol/L, higher than 1.7mmol/L is abnormal
Lipid profile index-LDL-C | baseline day 0, day 28
  LDL-C(Low-Density Lipoprotein Cholesterol) concentration level in the blood sample test: normal range 0-3.1mmol/L, higher than 3.1 mmol/L is abnomal;

SECONDARY OUTCOMES:
Number of AE and SAE | baseline day 0, through day 28
  The number of AE(Adverse Event) and SAE(Serious Adverse Event) associated with study product, reported during the trial period.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Cao, Principal Investigator — Jinhua Wenrong Hospital
Locations (2):
- China (2):
  - Raison Biotech Group Shanghai Lab, Shanghai, Shanghai Municipality
  - Jinhua Wenrong Hospital, Jinhua, Zhejiang

IPD SHARING:
Plan to Share IPD: No